CLINICAL TRIAL: NCT01812642
Title: A Double-Blind, Multiple Dose Titration Study to Investigate the Safety, Tolerability and Pharmacokinetics of Once Daily and Twice Daily Doses of JNJ-37822681 in Male and Female Patients With Stable Schizophrenia
Brief Title: A Pharmacokinetics Study to Evaluate Safety and Tolerability of JNJ-37822681 in Participants With Stable Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR014818; 2007-007669-20 (EudraCT Number); 37822681SCH2003
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; JNJ-37822681; Placebo
MeSH Terms: conditions — Schizophrenia | interventions — N-(1-(3,4-difluorobenzyl)piperidin-4-yl)-6-(trifluoromethyl)pyridazin-3-amine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- JNJ-37822681 10 milligram (Experimental): JNJ-37822681 oral capsule will be administered at a starting dose of 10 milligram (mg) twice daily for the first 3 days and thereafter dose will be titrated from Day 3 to Day 10 up to 80 mg per day and will be continued at same dose up to Day 14.
  Interventions: Drug: JNJ-37822681
- JNJ-37822681 20 milligram and placebo (Experimental): JNJ-37822681 oral capsule will be administered at a starting dose of 20 mg once daily for the first 3 days and thereafter dose will be titrated from Day 3 to Day 10 up to 80 mg per day and will be continued at same dose up to Day 14. Matching Placebo will be administered orally in the evening for 14 days (12 hour post JNJ-37822681 administration).
  Interventions: Drug: JNJ-37822681; Other: Placebo

INTERVENTIONS:
Drug: JNJ-37822681 — JNJ-37822681 oral capsule will be administered at a starting dose of either 20 mg (once daily) or 10 milligram (twice daily) for 14 days.
Other: Placebo — Matching Placebo will be administered orally, once daily in the evening (12 hour after JNJ-37822681 20 mg administration) for 14 days.
  Arms: JNJ-37822681 20 milligram and placebo

SUMMARY:
The purpose of this study is to evaluate safety, tolerability and pharmacokinetics (explores what the body does to the drug) of JNJ-37822681 in participants with stable schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self).

DETAILED DESCRIPTION:
This is a double-blind (neither physician nor participant knows the treatment that the participant receives), multi-center (conducted in more than one center), randomized (treatment group assigned by chance), and multiple-dose titration study of JNJ-37822681 in participants with stable schizophrenia. The total study duration will be approximately of 8 weeks per participant, consists of 4 parts: Screening (that is, 21 days before study commences on Day 1); Double-blind treatment (14 days); Follow-up (7 to 14 days after last dose administration). Participants will be randomly assigned to treatment with ascending dose levels of JNJ-37822681 once daily and twice daily. Efficacy will primarily be evaluated by Positive and Negative Syndrome Scale and Clinical Global Impression-Severity scale. Safety will be Barnes Akathisia Rating Scale, Abnormal Involuntary Movement Scale and Simpson Angus Rating Scale. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have schizophrenia diagnosis by Diagnostic and Statistical Manual of Mental Disorders, fourth edition (DSM-IV)
* known history of schizophrenia of at least 12 months by the referring psychiatrist
* Positive and Negative Syndrome Scale score at Screening less than 70
* Body Mass Index (BMI) between 18 and 35 kilogram divided by square meter inclusive (BMI =weight per square height)
* Female participants must meet any one of the following: postmenopausal (amenorrhea for at least 12 months and Follicle Stimulating Hormone levels of greater than 40 milli-international unit (MIU ) per milliliter at Screening), surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation or otherwise be incapable of pregnancy)

Exclusion Criteria:

* Any medical condition that could potentially alter the absorption, metabolism or excretion of the study medication, such as Crohn's (serious inflammation of any part of the gastrointestinal tract) disease, liver disease, or renal disease
* Relevant history of any significant and/or unstable cardiovascular, respiratory, neurologic (including seizures or significant cerebrovascular), renal, hepatic, endocrine or immunologic diseases
* History of neuroleptic malignant syndrome
* Female participants of childbearing potential
* Significant risk of suicidal or violent behavior

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score at Day 14 | Baseline and Day 14
  The AIMS rates the severity of involuntary movements from 0 (none) to 4 (severe), including facial and oral movements, extremity movements, trunk movements, global and judgments, and 2 additional items concerning dental status (yes/no). A total score (ranging from 0 to 28) will be calculated as the sum of items 1 to 7.
Barnes Akathisia Rating Scale (BARS) Score | Day 14
  The BARS includes an objective rating, 2 subjective ratings of symptoms of akathisia (awareness of restlessness and reported distress related to restlessness: range 0 to 3), and a global clinical rating of akathisia, ranging from 0 (absent) to 5 (severe). The global rating score, that is scored separately, is the most relevant measure of severity of akathisia. Higher scores denote worsening akathisia.
Change From Baseline in Simpson Angus Rating Scale (SAS) Score | Baseline and Day 14
  The SAS rates 10 items from 0 (normal) to 4 (extreme), including gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, leg pendulousness, head rotation, Glabellar tap, tremor and salivation. The SAS global score is the average score (total sum of items score divided by the number of items) and ranges between 0 and 4, where the higher score denotes more severe condition of extra pyramidal symptoms.

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) | 0 hour (Predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hour post administration of JNJ-37822681 on Day 1 and Day 14
  The Cmax is peak plasma concentration, determined by visual inspection of the data.
Concentration at Predose(Cpredose) | 0 hour (Predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hour post administration of JNJ-37822681 on Day 1 and Day 14
  Cpredose is predose plasma concentration (intermittent days and predose Day 14).
Average Concentration (Cavg) | 0 hour (Predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hour post administration of JNJ-37822681 on Day 1 and Day 14
  The Cavg is average plasma concentration at steady state and it will be calculated as AUC (τ)/τ (where time τ is the dosing interval).
Time to Reach Maximum Concentration(tmax) | 0 hour (Predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hour post administration of JNJ-37822681 on Day 1 and Day 14
  The Tmax is time to reach the peak plasma concentration and will be determined by visual inspection of the data.
Area Under the Plasma Concentration-Time Curve From 0 to 12 or 24 Hours Post Dosing (AUC 0-12h/24h) | 0 hour (Predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hour post administration of JNJ-37822681 on Day 1 and Day 14
  The AUC 0-12h/24h is area under the plasma concentration-time curve from 0 to 12 or from 0 to 24 hours post dosing on Day 1 and Day 14 and will be calculated by trapezoidal summation.
Area Under the Plasma Concentration-Time Curve From 0 to Tau Hours Post Dosing (AUC[0-tau]) | 0 hour (Predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 hour post administration of JNJ-37822681 on Day 1 and Day 14
  The AUC(0-tau) is area under the plasma concentration-time curve from 0 to τ hours post dosing at steady state and it will be calculated by trapezoidal summation (where time τ is the dosing interval).
Positive and Negative Syndromes Scale (PANSS) Total Score | Baseline up to 14 days after last study dose
  The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening.
Change From Baseline in Clinical Global Impression-Severity (CGI-S) Scale Score at Day 10 and 14 | Baseline, Day 10 and 14
  The CGI-S rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 is equivalent to "Normal, not at all ill" and a rating of 7 is equivalent to "Among the most extremely ill participants". Higher scores indicate worsening.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L.C Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (6):
- Antwerp, Belgium
- Germany (2):
  - Berlin
  - Neuss
- Nizny Novgorod, Russia
- Bratislava, Slovakia
- Stockholm, Sweden

REFERENCES:
- See also: A Double-Blind, Multiple Dose Titration Study to Investigate the Safety, Tolerability and Pharmacokinetics of Once Daily and Twice Daily Doses of JNJ-37822681 in Male and Female Patients With Stable Schizophrenia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=2181&filename=CR014818_CSR.pdf